CLINICAL TRIAL: NCT00664911
Title: Study of a Scale Predicting the Feasibility of Chemotherapy in Patients Aged 75 Years or Older With Solid Tumour
Brief Title: Combination Chemotherapy in Treating Older Patients With Solid Tumour,
Acronym: OLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDR0000593133; GERCOR-OLD; EudraCT-2007004103-36
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Solid Tumor Regardless of Localization and Stage
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Other): chemotherapy regimen
  Interventions: Other: chemotherapy

INTERVENTIONS:
Other: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This clinical trial is studying how well combination chemotherapy works in treating older patients with solid tumour.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine a prognostic scale of the feasibility of chemotherapy (at least two-thirds of the dose intensity usually administered) in patients aged 75 years or older with solid tumour.

Secondary

* To evaluate the efficacy, in terms of clinical and/or biological response, of treatments administered.
* To evaluate the incidence of severe (grade 3-4) toxicity.

OUTLINE: This is a multicenter study. Patients receive one of the following regimens according to cancer diagnosis and principal investigator preference. All regimens last 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumour regardless of localization or stage

PATIENT CHARACTERISTICS:

* > or = 75 years
* patient planned to receive > or = 2/3 of standard dose of the first cycle

PRIOR CONCURRENT THERAPY:

Chemonaive patient.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 516 (Actual)
Dates: Start 2008-03; Primary Completion 2012-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
chemotherapy feasibility | from inclusion to 3 months
  ability to deliver at least 3 months of the planned regimen therapy.
Number of patients receiving therapeutic dose-intensive therapy (doses must be at least equivalent to two-thirds the dose that is usually administered according to AMM recommendations) | 3 months
  dose reduction < 33%

SECONDARY OUTCOMES:
Grade 3-4 toxicities according to NCI-CTCAE version 3 | from inclusion to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Carola, MD, Study Chair — C.H. Senlis
Locations (29):
- France (29):
  - Centre Radiotherapie Oncologie Moyenne Garonne, Agen
  - Centre Hospitalier de Castelluccio, Ajaccio
  - Centre Hospitalier d'Ardeche Meridionale, Aubenas
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - Centre Hospitalier de Beauvais, Beauvais
  - Clinique des Cedres, Cornebarrieu
  - Centre Medico-Chirurgical et Obstetrique d'Evry, Évry
  - Hopital Clarac, Fort de France Cedex
  - Centre Hospitalier Intercommunal des Alpes du Sud, Gap
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Centre Hospitalier St. Joseph St. Luc, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Hospitalier Chanaux, Mâcon
  - Centre Hospitalier de Montelimar, Montélimar
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital de la Croix St. Simon, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital Rene Dubos, Pontoise
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Prive Saint-Gregoire, Saint-Grégoire
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Centre Hospitalier de Semur en Auxois, Semur-en-Auxois
  - C.H. Senlis, Senlis
  - Hopital Foch, Suresnes
  - Centre hospitalier de Tonnerre, Tonnerre
  - Centre Hospitalier Villeneuve Saint Georges, Villeneuve-Saint-Georges